CLINICAL TRIAL: NCT04289207
Title: Phase II Trial of Romiplostim With Danazol in Patients With Eltrombopag-resistant Immune Thrombocytopenia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Kyowa Kirin Korea Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Youngil Koh, Associate professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0620200130
Record Dates: First submitted 2020-02-25; First posted 2020-02-28 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — romiplostim; Danazol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Romiplostim and danazol (Experimental): Treatment group (romiplostim and danazol)
  Interventions: Drug: Romiplostim and danazol

INTERVENTIONS:
Drug: Romiplostim and danazol — Treatment with romiplostim and danazol

SUMMARY:
In this study, we tried to demonstrate clinical benefit of additive danazol to romiplostim therapy in patients with eltrombopag-resistant immune thrombocytopenia

DETAILED DESCRIPTION:
The patients with eltrombopag-resistant immune thrombocytopenia are treated with romiplostim and danazol. The efficacy and toxicity of treatment will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* aged over 18 years
* diagnosed with immune thrombocytopenia (bone marrow examination is not necessary)
* failed to achieve platelet count over 50X10^9/L with eltrombopag
* ECOG performance status 0,1,2
* available to obtain informed consent

Exclusion Criteria:

* Hepatitis B or C carriers
* HIV positive patients
* diagnosed with systemic lupus erythematosus or other autoimmune disorders
* unable to intake orally or absorb through gastrointestinal tract
* pregnant or breast-feeding
* diagnosed with uncontrolled seizure or other neuropsychiatric disorders
* diagnosed with clinically significant cardiovascular events within 6 months or dyspnea on exertion evaluated to New York Heart Association Functional Classification III or IV
* diagnosed with clinically significant cerebrovascular disorders
* previously diagnosed or treated with thromboembolism
* current treating malignant diseases
* currently accompanied by uncontrolled infection or active bleeding
* with blood test results as follows; total bilirubin > 2xUNL(upper normal limit), AST/ALT > 1.5xUNL, creatinine > 1.5xUNL, glomerular filtration rate < 30ml/min/1.73m^2
* registered to other clinical trials for treatment of immune thrombocytopenia
* judged to be inappropriate for clinical trial by doctor in charge

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Response rate | week 8
  proportion of patients with platelet count over 50x10^9/L

SECONDARY OUTCOMES:
Time to best response | week 24
  time interval between initiation of treatment and best response
Response duration | week 24
  period of time with platelet count over 50x10^9/L
Effects on quality of life | week 24
  changes in EORTC QLQ-C30 scores

CONTACTS AND LOCATIONS:
Overall Officials: Youngil Koh, Principal Investigator — Seoul National University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cooper N, Bussel J. The pathogenesis of immune thrombocytopaenic purpura. Br J Haematol. 2006 May;133(4):364-74. doi: 10.1111/j.1365-2141.2006.06024.x. PMID 16643442
- [Background] Bussel JB, Kuter DJ, Pullarkat V, Lyons RM, Guo M, Nichol JL. Safety and efficacy of long-term treatment with romiplostim in thrombocytopenic patients with chronic ITP. Blood. 2009 Mar 5;113(10):2161-71. doi: 10.1182/blood-2008-04-150078. Epub 2008 Nov 3. PMID 18981291
- [Background] Wong RSM, Saleh MN, Khelif A, Salama A, Portella MSO, Burgess P, Bussel JB. Safety and efficacy of long-term treatment of chronic/persistent ITP with eltrombopag: final results of the EXTEND study. Blood. 2017 Dec 7;130(23):2527-2536. doi: 10.1182/blood-2017-04-748707. Epub 2017 Oct 17. PMID 29042367
- [Background] Khellaf M, Viallard JF, Hamidou M, Cheze S, Roudot-Thoraval F, Lefrere F, Fain O, Audia S, Abgrall JF, Michot JM, Dauriac C, Lefort S, Gyan E, Niault M, Durand JM, Languille L, Boutboul D, Bierling P, Michel M, Godeau B. A retrospective pilot evaluation of switching thrombopoietic receptor-agonists in immune thrombocytopenia. Haematologica. 2013 Jun;98(6):881-7. doi: 10.3324/haematol.2012.074633. Epub 2013 Feb 26. PMID 23445876